CLINICAL TRIAL: NCT07404397
Title: Comparing Adjuvant Treatments for High Tone Pelvic Floor Dysfunction: a Pilot Randomized Controlled Trial
Brief Title: Comparing Adjuvant Treatments for High Tone Pelvic Floor Dysfunction
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The American Association of Obstetricians and Gynecologists Foundation (Unknown)
Responsible Party: Principal Investigator, Sara Till, MD, MPH, Assistant Professor of Obstetrics and Gynecology, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00280388
Record Dates: First submitted 2026-02-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: High Tone Pelvic Floor Dysfunction
Keywords: pelvic floor physical therapy; cyclobenzaprine; vibrating pelvic floor massage wand
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cyclobenzaprine PFPT (Experimental): During Phase 1, participants will be instructed to use cyclobenzaprine as detailed below. During Phase 2, participants will complete a course of pelvic floor physical therapy and will continue using cyclobenzaprine.
  Interventions: Drug: Cyclobenzaprine; Procedure: Pelvic floor physical therapy
- Pelvic floor massage wand & PFPT (Experimental): During Phase 1, participants will be instructed to use pelvic floor massage wand as detailed below. During Phase 2, participants will complete a course of pelvic floor physical therapy and will continue using pelvic floor massage wand.
  Interventions: Device: Pelvic floor massage wand; Procedure: Pelvic floor physical therapy

INTERVENTIONS:
Drug: Cyclobenzaprine — Participants will be instructed to use cyclobenzaprine IR 5mg at bedtime. We will encourage participants to take the medication in the evening/before bed to minimize potential for bothersome sedation. Participants will be given the option to begin with ½ tablet (2.5mg) if preferred and titrate to 5mg dose, with goal of minimizing sedation side effects. Participants will be instructed that they may increase to 10mg at bedtime at Day 14 if desired based on perceived benefits and side effects.
  Other Names: Flexeril
  Arms: Cyclobenzaprine PFPT
Device: Pelvic floor massage wand — Participants will be instructed to use a commercially available vibrating pelvic floor massage wand for approximately 10-15 minutes at least 3 times per week, which can be titrated as needed (standard use recommendations per our pelvic physical therapists).
  Arms: Pelvic floor massage wand & PFPT
Procedure: Pelvic floor physical therapy — Pelvic floor physical therapy for HTPFD uses manual manipulation to release localized muscle tension or trigger points, improve mobility of fascia, and address orthopaedic issues such as pelvic alignment and spine/hip mobility to reduce pain and improve function.

SUMMARY:
The researchers are comparing two treatments for high tone pelvic floor dysfunction (HTPFD) in conjunction with pelvic floor physical therapy (PFPT). The goal of this study is to find out which of two extra treatments works better for people with HTPFD when they also do regular PFPT. First, the researchers will compare a muscle relaxant medicine (cyclobenzaprine IR) to using a vibrating pelvic floor massage wand. Everyone in the study will also do pelvic floor physical therapy. The researchers want to see how these treatments affect pain, sexual health, physical ability, and overall quality of life.

DETAILED DESCRIPTION:
Devices such as the Intimate Rose Vibrating Pelvic Floor Massage Wand are not required to indicate a phase for ClinicalTrials.gov. However, this study is marked as phase 2/3 considering the use of a study drug, Cyclobenzaprine.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported moderate to severe chronic pelvic pain for >6 months duration at time of screening visit. Moderate to severe chronic pain is defined as >4 on 0-10 (worst daily pain) for >14 days per month. Pelvic pain is defined as pain perceived to be located in the anatomic pelvis.
* Diagnosis of high tone pelvic floor dysfunction (HTPFD), defined as >12/60 summative pelvic floor tenderness score on standardized pelvic examination by chronic pelvic pain specialist (MD or NP) within the past year
* Referred to pelvic floor physical therapy (PFPT) by their chronic pelvic pain specialist for management of HTPFD
* Willing to undergo a 12-session course of PFPT for HTPFD, including internal/vaginal tissue manipulation per standardized protocol
* Willing to delay start of PFPT until Phase 2 of the trial
* Willing to be randomized to either daily use of cyclobenzaprine or use of vibrating pelvic floor muscle massage wand for total of 18 weeks
* Willing to undergo standardized pelvic floor myofascial exam three times over the study period (baseline, end of Phase 1, end of Phase 2)
* Willing to undergo quantitative sensory testing (QST) two times over the study period (baseline, end of Phase 1)
* Willing to undergo blood draw two times over the study period (baseline, end of Phase 1)
* Ability to read and speak English to allow for written informed consent, phenotyping, and patient-reported outcome measures
* No plans for pregnancy within the next 12 months

Exclusion Criteria:

* Hypersensitivity or allergy to cyclobenzaprine or any component of cyclobenzaprine
* Underwent PFPT within 6 months of screening date
* Pregnancy at any point during study period (self-reported home urine pregnancy test or serum b-Hcg test, positive urine pregnancy test at baseline, post-Phase 1, or post-Phase 2 study visits).
* Currently breastfeeding at time of screening visit
* Scheduled for or are planning moderate/major gynecologic surgery (including hysterectomy, excision of endometriosis, ovarian cystectomy/oopherectomy, myomectomy) within the following 6 months of screening date
* Current (at time of screening visit) diagnosis of postural orthostatic tachycardia syndrome
* Current significant neurologic or musculoskeletal conditions that would preclude participation in PFPT (cerebral palsy, severe hip/back osteoarthritis that would prevent lithotomy position during sessions)
* Unwilling to avoid or stop baseline use of cyclobenzaprine and other muscle relaxants (including methocarbamol, tizanidine, baclofen, carisoprodol, metaxalone)
* Current use of tricyclic antidepressants
* Current use of monoamine oxidase inhibitor
* Current use of vaginally delivered benzodiazepine such as diazepam (more than once per month) and unwilling to stop use of vaginally delivered benzodiazepine for the duration of this study
* Current diagnosis of hyperthyroidism
* Current diagnosis of moderate or severe hepatic impairment
* Myocardial infarction within prior 12 months
* Current diagnosis of congestive heart failure
* Current cardiac pacemaker in place
* Current diagnosis of closed angle glaucoma
* Current major psychiatric condition (including psychosis or suicidal ideation within past year)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference 4a score | Baseline, 18 weeks
  PROMIS pain interference 4a score is from 4 questions with score ranging from 4-20. Higher scores indicate greater pain interference
PROMIS pain interference 4a score | Baseline, 6 weeks
  PROMIS pain interference 4a score is from 4 questions with score ranging from 4-20. Higher scores indicate greater pain interference

SECONDARY OUTCOMES:
50% reduction in PROMIS pain interference 4a score | 18 weeks compared to baseline
  PROMIS pain interference 4a score is from 4 questions with score ranging from 4-20. Higher scores indicate greater pain interference
PROMIS pain intensity 1a score | Baseline, 18 weeks
  PROMIS pain intensity 1a score is 1 question ranging from 0-10 and the higher the number the worse the pain.
PROMIS pain intensity 1a score | Baseline, 6 weeks
  PROMIS pain intensity 1a score is 1 question ranging from 0-10 and the higher the number the worse the pain.
Female Sexual Function Index (FSFI) | Baseline, 18 weeks
  Female Sexual Function Index (FSFI) overall score has six domains and a maximum score of 36, with a higher score indicating better functioning.
Female Sexual Function Index (FSFI) | Baseline, 6 weeks
  Female Sexual Function Index (FSFI) overall score has six domains and a maximum score of 36, with a higher score indicating better functioning.
PROMIS Self Efficacy for Managing Symptoms SF 4a | Baseline, 18 weeks
  PROMIS Self Efficacy for Managing Symptoms SF 4a is 4 questions with scores ranging from 4-20. Highter scores indicate higher confidence in symptom management
PROMIS Self Efficacy for Managing Symptoms SF 4a | Baseline, 6 weeks
  PROMIS Self Efficacy for Managing Symptoms SF 4a is 4 questions with scores ranging from 4-20. Highter scores indicate higher confidence in symptom management
Summative pelvic floor myofascial tenderness to palpation | Baseline, 18 weeks
  For Bilateral pubococcygeus, Bilateral iliococcygeus, and Bilateral obturator internus
Summative pelvic floor myofascial tenderness to palpation | Baseline, 6 weeks
  For Bilateral pubococcygeus, Bilateral iliococcygeus, and Bilateral obturator internus
Patient Global Impression of Change | 18 weeks
  The Patient Global Impression of Change is scored on a scale of 1 - 7, with a score of 1 representing that the patient was very much worse following the trial, and a score of 7 representing that the patient was very much improved following the course of the trial.
Patient Global Impression of Change | 6 weeks
  The Patient Global Impression of Change is scored on a scale of 1 - 7, with a score of 1 representing that the patient was very much worse following the trial, and a score of 7 representing that the patient was very much improved following the course of the trial.
Number of pelvic floor physical therapy (PFPT) sessions attended | Up to 18 weeks
  PFPT session attendance will be tracked by patient self-report

CONTACTS AND LOCATIONS:
Overall Officials: Sara Till, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified, anonymized data sets underlying all publications resulting from the proposed research involving human subjects will be shared with legitimate academic researchers and other community members with a legitimate scientific interest in the research. Where practicable, sharing will take place under a written agreement between the principal investigators prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the datasets. The aim is to permit others to validate and replicate research findings described in the Aims while protecting participant confidentiality.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The research community will have access to the data when the award ends.
Access Criteria: academic researchers and other community members with a legitimate scientific interest in the research. Members of the scientific community who would like a curated copy of the final datasets (i.e., datasets underlying publications) from this study can request a copy by contacting the principal investigators.